CLINICAL TRIAL: NCT05645484
Title: The Prognostic Value of 18F-PFPN PET Imaging in Patients With Malignant Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: XLan-0624
Record Dates: First submitted 2022-12-02; First posted 2022-12-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18F-PFPN PET imaging: For clinically suspected or confirmed melanoma patients, targeted melanin-specific imaging 18F-PFPN PET/MR was performed. CT was instead when MRI was contraindicated. PET images, clinical characteristics, and follow-up information will be collected for prognostic analyses.
  Interventions: Drug: 18F-PFPN
- 18F-FDG PET imaging: For clinically suspected or confirmed melanoma patients, general metabolic imaging 18F-FDG PET PET/CT was performed. PET images, clinical characteristics, and follow-up information will be collected for prognostic analyses.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-PFPN — 18F-PFPN (dose: 3.0-5.4 MBq/kg) will be injected intravenously prior to imaging.
  Other Names: 18F-PEG3-FPN
  Groups: 18F-PFPN PET imaging
Drug: 18F-FDG — 18F-FDG (dose: 3.7-5.4 MBq/kg) will be injected intravenously prior to imaging.
  Other Names: 18F-fluorodeoxyglucose
  Groups: 18F-FDG PET imaging

SUMMARY:
This is a monocentric prospective study. This study aims to investigate the prognostic value of the novel melanin-targeted imaging modality 18F-PFPN PET in patients with melanoma and seek independent prognostic factors for progression-free survival (PFS) and overall survival (OS). The patients with clinically highly suspected or confirmed melanoma who underwent 18F-PFPN and 18F-FDG PET scans will be enrolled consecutively. Patients' PET images, clinical characteristics, and follow-up information will be collected for prognostic analyses. This study plans to set the sample size as 100 cases.

DETAILED DESCRIPTION:
Melanoma is an aggressive malignancy with a high mortality rate. Accurate diagnosis and prognostic risk assessment are essential to the clinical management of melanoma. Melanin is present in most melanoma and has become a potential target for melanoma. This team has successfully synthesized a positron nuclide targeting melanin probe named 18F-PFPN (18F-N-(2-diethylaminoethyl)-4-(2-[2-ethoxy]-ethoxy) pyridine), which has been proven to be safe and well-tolerated. It has shown excellent diagnostic value in both primary and metastatic melanoma. This prospective study was designed to further investigate the prognostic value of 18F-PFPN for melanoma and compare it with the general metabolic imaging agent 18F-FDG. In this study, patients with clinically highly suspected or confirmed melanoma who underwent 18F-PFPN and 18F-FDG PET scans will be enrolled consecutively. Patients' PET images, clinical characteristics, and follow-up information will be collected for prognostic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically confirmed melanoma;
* Patients with complete clinical and follow-up data (including TNM stage, subtypes, and treatment strategies).

Exclusion Criteria:

* Uncertain histopathology;
* A history of other malignancies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically highly suspected or confirmed melanoma underwent 18F-PFPN and 18F-FDG PET scans in the PET center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 1-2 years
  PFS time is calculated from the date of PET imaging to the first recurrence/progression or death or the endpoint of follow-up. The disease recurrence/progression is confirmed after a thorough review of following-up imaging or pathologic findings.
Overall Survival (OS) | 1-2 years
  OS time is defined as the time from PET imaging to death or the endpoint of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhang X, Lin Z, Li M, Gai Y, Zheng H, Fan L, Ruan W, Hu F, Chen J, Lan X. Melanin-targeted [18F]-PFPN PET imaging for prognosticating patients with melanoma. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):3062-3071. doi: 10.1007/s00259-023-06258-5. Epub 2023 May 16. PMID 37191681